CLINICAL TRIAL: NCT05325437
Title: The Effect of Laparoscopic Splenectomy and Azygoportal Disconnection on Liver Reserve Function for Cirrhosis Patients
Acronym: ELSDL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Guo-Qing Jiang, Clinical Professor, Northern Jiangsu People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YZUC-007
Record Dates: First submitted 2022-03-18; First posted 2022-04-13 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Cirrhosis, Liver; Splenectomy; Status; Portal Hypertension
Keywords: Cirrhosis; Splenectomy; Azygoportal disconnection; Laparoscopy; Liver Reserve Function
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Laparoscopic splenectomy and azygoportal disconnection
  Interventions: Procedure: Laparoscopic splenectomy and azygoportal disconnection

INTERVENTIONS:
Procedure: Laparoscopic splenectomy and azygoportal disconnection — The laparoscopic splenectomy and azygoportal disconnection was performed by the same surgical team.

SUMMARY:
In this study, the investigators compared the improvement of liver reserve function related indicators in patients with liver cirrhosis after laparoscopic splenectomy and azygoportal disconnection. To determine whether surgical treatment can help enhance postoperative liver reserve function and improve patient prognosis.

DETAILED DESCRIPTION:
The patients were enrolled according to the research criteria, and collected the general basic information of the patients. After the preoperative preparation was perfected, the same surgical team performed laparoscopic splenectomy and azygoportal disconnection, and the same nursing team performed the nursing after the operation. Then, patients received a unified treatment plan after surgery, including medication, other treatments and follow-up. During the treatment, the liver reserve function related indicators of the patients were monitored before surgery, 3, 6, 12 and 24 months after surgery, including TBIL, DBIL, ALB, ALT, INR, PT, Child-Pugh, ascites, prealbumin, ICG-K, ICG-R 15 and ICG-T/2.

ELIGIBILITY:
Inclusion Criteria:

* A clinical, radiological or histologic diagnosis of cirrhosis of any etiology
* Splenomegaly with secondary hypersplenism
* gastroesophageal variceal bleeding
* Informed consent to participate in the study

Exclusion Criteria:

* Hepatocellular carcinoma or any other malignancy,
* Child-Pugh grade C
* Recent peptic ulcer disease
* History of Hemorrhagic stroke
* Pregnancy.
* Uncontrolled Hypertension
* Human immunodeficiency virus (HIV) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Liver reserve function ICG-K at 3 months after surgery. | 3 months
  The level of liver reserve function ICG-K at 3 months after surgery.
Liver reserve function ICG-K at 6 months after surgery. | 6 months
  The level of liver reserve function ICG-K at 6 months after surgery.
Liver reserve function ICG-K at 12 months after surgery. | 12 months
  The level of liver reserve function ICG-K at 12 months after surgery.
Liver reserve function ICG-K at 24 months after surgery. | 24 months
  The level of liver reserve function ICG-K at 24 months after surgery.
Liver reserve function ICG-R 15 at 3 months after surgery. | 3 months
  The level of liver reserve function ICG-R 15 at 3 months after surgery.
Liver reserve function ICG-R 15 at 6 months after surgery. | 6 months
  The level of liver reserve function ICG-R 15 at 6 months after surgery.
Liver reserve function ICG-R 15 at 12 months after surgery. | 12 months
  The level of liver reserve function ICG-R 15 at 12 months after surgery.
Liver reserve function ICG-R 15 at 24 months after surgery. | 24 months
  The level of liver reserve function ICG-R 15 at 24 months after surgery.
Liver reserve function ICG-T/2 at 3 months after surgery. | 3 months
  The level of liver reserve function ICG-T/2 at 3 months after surgery.
Liver reserve function ICG-T/2 at 6 months after surgery. | 6 months
  The level of liver reserve function ICG-T/2 at 6 months after surgery.
Liver reserve function ICG-T/2 at 12 months after surgery. | 12 months
  The level of liver reserve function ICG-T/2 at 12 months after surgery.
Liver reserve function ICG-T/2 at 24 months after surgery. | 24 months
  The level of liver reserve function ICG-T/2 at 24 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Guo-Qing Jiang, MD, Study Chair — Clinical Medical College of Yangzhou University
Locations (1):
- Clinical Medical College of Yangzhou University, Yangzhou, Jiangsu, China